CLINICAL TRIAL: NCT03489824
Title: The Effectiveness of Right- vs Left-lateral Starting Position in Unsedated Colonoscopy With Modified-Water Immersion Method Colonoscopy
Brief Title: Effectiveness of RL- vs LL-starting Position in Unsedated Water Immersion Colonoscopy
Acronym: RLPvsLLP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, PUTUT BAYUPURNAMA, MD, Internist-Gastroenterohepatology Consultant, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PB-WC003
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Water Immersion Method Colonoscopy in Unsedated Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified-WIM colonoscopy in RLP (Experimental): Modified-water immersion method colonoscopy is performed to patients with right-lateral starting position (RLP). Patients will lie in the right lateral position with both hips and knees flexed at the beginning and change the position into supine and at last left-lateral position when it is needed.
  Interventions: Procedure: modified- WIM colonoscopy
- modified-WIM colonoscopy in LLP (Active Comparator): Modified-water immersion method (WIM) colonoscopy is performed to patients with left-lateral starting position (LLP). Patients will lie in the left lateral position with right hip and knee flexed and left leg straight at the beginning and change the position into supine and at last right lateral position when it is needed.
  Interventions: Procedure: modified- WIM colonoscopy

INTERVENTIONS:
Procedure: modified- WIM colonoscopy — Modified-water immersion method of colonoscopy refers to the freely episodic suction of the infused-water during colonoscopy insertion phase at a moment to negotiate the angulated colon to facilitate cecal intubation but not suction the mucosa. The original water immersion method only suctions the water when the colon is over-distended or it is dirty and exchanges it with the new cleans water during insertion then evacuates all of the water during withdrawal
  Other Names: modified-water immersion method colonoscopy

SUMMARY:
Abdominal discomfort is of the most important patient interest when in an unsedated colonoscopy examination. Water method for colonoscopy examination has been studied widely and evidence showed effectiveness in reducing discomfort and increase cecal intubation time and increasing cecal intubation rates in unsedated patients.

DETAILED DESCRIPTION:
Abdominal discomfort is of the most important patient interest when in an unsedated colonoscopy examination. Water method for colonoscopy examination has been studied widely and evidence showed effectiveness in reducing discomfort and increase cecal intubation time and increasing cecal intubation rates in unsedated patients. Our previous studies showed that water immersion method reduced the VAS score, accelerated the intubation time significantly without different changing cecal intubation rate. Previous right-sided vs. left-sided starting position colonoscopy study in sedated patients with air insufflation colonoscopy method showed that right-sided starting position improved the abdominal discomfort score and faster cecal intubation time. We want postulate that the right-sided starting position can also maximize the water method advantages in lowering the discomfort score, faster cecal intubation time and higher cecal intubation rates, and it will improve patient acceptance of water unsedated colonoscopy and willingness to repeat.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years old with the indication for colonoscopy, such as chronic diarrhea, chronic constipation, hematochezia, chronic lower abdominal pain, positive fecal occult blood test, and other change of bowel habit symptoms indicative of the need for diagnostic colonoscopy examination.

Exclusion Criteria:

* Patients who refuse to participate, patients with obstructive lesions in the colon distal of the cecum. , patients with experienced colon resection, patients who are hemodynamically unstable, and patients with severe cardiac disorders (such as acute myocardial infarction, unstable angina, malignant arrhythmia, and moderate to severe congestive heart failure ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Abdominal discomfort score | during the study
  The patient reported level of abdominal discomfort experienced during the colonoscopy examination. The patients will punctuate the VAS score line form by themselves, immediately after the end of examination (patient still lying on the examination bed). The VAS will be measured on a linear visual analog scale: 0=none, 10=most severe.

SECONDARY OUTCOMES:
Cecal Intubation rate | during the study
  The proportion of patients with successful insertion of the colonoscope to the cecum with the tip of the colonoscope touching the floor of the cecum with visualization of the medial cecal wall between the ileocecal valve and/or appendix orifice
Cecal intubation time | during the study
  Time need to insert from the anus to the cecum
Time needs to pass rectosigmoid | during the study
  Time needs to pass rectosigmoid is measured from the insertion until to when the colonoscope length passes the 40 cm sign on the colonoscope without looping.
Difficulties during colonoscope insertion | during the study
  Difficulties which are found during colonoscope insertion will be recorded and analyzed (e.g., looping; predominant faecal obstruction visualization level, need to use abdominal compression, need to change from starting position)

OTHER OUTCOMES:
Willingness to repeat the colonoscopy examination | during the study
  0=No or 1=Yes, patient fill the questionnaire form by themselves

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Room of Dr Sardjito General Hospital, Yogyakarta, Special Province of Yogyakarta, Indonesia

REFERENCES:
- [Derived] Bayupurnama P, Ratnasari N, Indrarti F, Triwikatmani C, Maduseno S, Nurdjanah S, W Leung F. The Effectiveness of Right- vs Left-lateral Starting Position in Unsedated Diagnostic Colonoscopy with Modified-water Immersion Method: A Randomized Controlled Trial Study. Clin Exp Gastroenterol. 2020 Sep 24;13:369-375. doi: 10.2147/CEG.S270793. eCollection 2020. PMID 33061515